CLINICAL TRIAL: NCT01716377
Title: Healing With Venlafaxine After Injury: A Randomized Clinical Trial of Venlafaxine Following Motor Vehicle Collision
Brief Title: Healing With Venlafaxine After Injury (HELP)
Acronym: HELP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Mayday Fund (Other); University of North Carolina (Other); University of Cincinnati (Other); Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Francesca Beaudoin, Assistant Professor of Emergency Medicine, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 104106
Record Dates: First submitted 2012-10-25; First posted 2012-10-29 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Neck Pain
Keywords: Neck Pain; Musculoskeletal pain; Venlafaxine
MeSH Terms: conditions — Neck Pain; Musculoskeletal Pain | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 37.5mg QD 1 week 75mg QD 1 week 150mg QD 8 weeks 75mg QD 1 week 37.5mg QD 1 week
  Interventions: Drug: Venlafaxine
- Venlafaxine (Active Comparator): 37.5mg QD 1 week 75mg QD 1 week 150mg QD 8 weeks 75mg QD 1 week 37.5mg QD 1 week
  Interventions: Drug: Venlafaxine

INTERVENTIONS:
Drug: Venlafaxine — Sixty patients who present following a minor motor vehicle collision will be randomized to venlafaxine vs. placebo, and the ability of venlafaxine to decrease acute and persistent musculoskeletal neck pain will be assessed.
  Other Names: Effexor

SUMMARY:
Purpose: The purpose of this study is to demonstrate the potential efficacy of venlafaxine administration in reducing acute and chronic musculoskeletal pain in individuals presenting to the ED for evaluation after motor vehicle collision.

Participants: Participants will consist of 60 patients between the ages of 18-50 who present to the ED within 12 hours post-motor vehicle collision. Patients who report a neck pain score > 6 will be screened for further eligibility.

Procedures (methods): Using a placebo-controlled, randomized, double-blind trial design, 60 high risk patients will be randomized to venlafaxine vs. placebo in the ED. The ability of venlafaxine to decrease acute and persistent musculoskeletal neck pain will be assessed during serial short-term telephone follow-ups as well as more in-depth follow-ups at 6 weeks, 4 months, and 6 months post-MVC.

DETAILED DESCRIPTION:
Results from both animal and human studies suggest that treatment with the serotonin-norepinephrine reuptake inhibitor (SNRIs) venlafaxine may reduce post-MVC pain. In addition, venlafaxine has been shown to be beneficial in reducing posttraumatic stress disorder (PTSD) symptoms, and in some patients PTSD symptoms may contribute to reinforcing pain persistence after trauma.

This phase IIB pilot trial will screen patients presenting to the ED after MVC for the presence of severe axial pain (>4 on a 0-10 numeric rating scale). Sixty of these "high risk" patients will be randomized to venlafaxine vs. placebo, and the ability of venlafaxine to decrease acute and persistent musculoskeletal axial pain will be assessed.

Results will be used to design a large-scale RCT assessing the efficacy of venlafaxine intervention in decreasing acute and persistent musculoskeletal pain in high-risk patients presenting to the ED after minor MVC.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 59
* Presents to ED within 24 hours of MVC
* ED axial pain score greater than or equal to 4 (0-10 NRS)
* Clinically sober
* Willing to provide a blood sample
* Has a telephone
* Has regular access to Internet and an email address
* Able to speak and read English
* Permanent US citizen or has a green card
* Blood pressure reading(s) in ED that, when considered in the context of patient past and current history, in the investigator's judgment does not exceed acceptable level

Exclusion Criteria:

* Axial pain score greater than 0 in the past month (0-10 NRS)
* Clinically unstable
* Fracture (other than fracture of the phalanges)
* Substantial soft tissue injury
* Hepatic failure (acute or chronic)
* Renal failure (acute or chronic)
* Coronary artery disease, including previous MI, Angina, PCTA, etc.
* History of glaucoma
* Previous congestive heart failure
* History of seizure disorder
* History of mania or psychotic disorder
* History of suicidal ideation
* Prisoner
* History and behavior indicates, in the investigator's judgment, that the participant would likely be noncompliant with the study
* Any other condition that, in the investigator's judgment, would indicate that the patient in unsuitable for the study (e.g. might interfere with the study, confound interpretation, or endanger patient)
* Currently taking a monoamine oxidase inhibitor
* Currently taking medication with substantial interaction with venlafaxine, or which could confound interpretation of study results
* Breastfeeding
* If female, either not postmenopausal (having menses within past year), or, if childbearing potential, positive pregnancy test prior to randomization and not using a medically acceptable form of contraception
* Exceeds acceptable chronic daily opioid use prior to MVC
* Previously on venlafaxine
* Previous allergic reaction to venlafaxine
* Antidepressant use within 2 weeks of study start (4 week if Prozac)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Average neck pain | 0-31 Days
  The primary outcome variable is average neck pain (0 - 10 numeric rating pain score recorded from patient) after study drug initiation through Day 31.

SECONDARY OUTCOMES:
Chronic neck pain | Study day 38 through 6 months
  The secondary outcome variable is average neck pain (0 - 10 numeric rating pain score recorded from patient) between study day 38 through 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel A McLean, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill; Jeffrey Jones, MD, Principal Investigator — Corewell Health West; Kirsten Rindal, MD, Principal Investigator — University of Rochester; Gregory Fermann, MD, Principal Investigator — University of Cincinnati
Locations (3):
- United States (3):
  - Spectrum Health, Grand Rapids, Michigan
  - University of Rochester Medical Center, Rochester, New York
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No